CLINICAL TRIAL: NCT04017793
Title: The Neural Changes Associated With a Mindfulness Intervention for Adults With Autism Spectrum Disorder
Brief Title: Mindfulness-Associated Brain Changes in Adults With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Southwest Autism Research and Resource Center (SARRC) (Unknown); Banner Alzheimer's Institute (Other)
Responsible Party: Principal Investigator, Brittany Blair Braden, Assistant Professor; Autism and Brain Aging Laboratory Director, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB # STUDY00007227
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Stress Reduction Program (Active Comparator)
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Relaxation Group (Active Comparator)
  Interventions: Behavioral: Relaxation Group

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — Structured 8-week training program teaching about increased mindfulness strategies and gentle stretching.
  Arms: Mindfulness Based Stress Reduction Program
Behavioral: Relaxation Group — 8-weekly group discussion meetings reviewing relaxation techniques and other stress reduction strategies with an emphasis on social support.
  Arms: Relaxation Group

SUMMARY:
The purpose of this study to measure brain functioning before and after stress-reduction classes to better understand how symptom improvements relate to brain functioning in adults with ASD (Autism Spectrum Disorder). Participants will be randomly assigned to one of two stress reduction classes that will meet once a week for 8 weeks. One group will complete a structured training program called Mindfulness Based Stress Reduction (MBSR) that involves teaching about increased mindfulness strategies and gentle stretching. The other group will review relaxation techniques and other stress reduction strategies and will include social support. Structural and functional MRI, EEG, and behavioral self-report data will be collected to understand more about how the brain changes in subtle ways when people feel better and are more aware of their emotional state.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 89 years old, with a special focus on adults with ASD who are going to college given the additional stress of this phase in life. We are recruiting participants across a broad age range in order to maximize our ability to inform interventions for adults with ASD. The upper age limit of 89 years was selected so a de-identified dataset can be created with all participant ages included.
* ASD diagnosis via gold-standard diagnostic assessments (Autism Diagnostic Observation Schedule-2).
* Must be able to attend at least 7 of the 8 weekly intervention classes.
* English speaking: Participants must be English-speaking because the screening and behavioral measures are in English (including the intelligence estimate).

Exclusion Criteria:

* Participants with Intelligence Quotient (IQ) scores <70 will be excluded to minimize variability due to general cognitive functioning.
* Report of any major medical illnesses, histories of seizures, or head trauma with loss of consciousness. These health factors can cause brain changes that would confound findings.
* Concerns that the participant may not be able to complete the MRI neuroimaging requirements for the study, including claustrophobia or metal objects within the participant's body or eyes. Implanted metal objects may create a safety hazard in the powerful magnetic field during MRI imaging.
* Pregnant women. MRI has no known effects on pregnancy or fertility. However, since we are not 100% certain MRI has no effects on a developing fetus, women who are pregnant may not participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory - II | Baseline; Pre-intervention
  21-question multiple-choice self-report inventory for measuring depression severity. Items are rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63. Raw scores ranging from 0-13 indicate minimal depression. Raw scores ranging from 14-19 indicate mild depression. Raw scores of 20-28 indicate moderate depression and scores of 29-63 indicate severe depression.
Beck Depression Inventory - 2 | Post-intervention (~10 weeks)
  21-question multiple-choice self-report inventory for measuring depression severity. Items are rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63. Raw scores ranging from 0-13 indicate minimal depression. Raw scores ranging from 14-19 indicate mild depression. Raw scores of 20-28 indicate moderate depression and scores of 29-63 indicate severe depression.
State-Trait Anxiety Inventory | Baseline; Pre-intervention
  Self-report inventory measuring two types of anxiety. 20 items assess the temporary condition of state anxiety, or anxiety about an event, and an additional 20 items assess the more general trait anxiety, or anxiety level as a personal characteristic. Items are rated on a 4-point frequency scale. Scores range from 20 to 80, with higher scores correlating with greater anxiety.
State-Trait Anxiety Inventory | Post-intervention (~10 weeks)
  Self-report inventory measuring two types of anxiety. 20 items assess the temporary condition of state anxiety, or anxiety about an event, and an additional 20 items assess the more general trait anxiety, or anxiety level as a personal characteristic. Items are rated on a 4-point frequency scale. Scores range from 20 to 80, with higher scores correlating with greater anxiety.

SECONDARY OUTCOMES:
World Health Organization Quality of Life | Baseline; Pre-intervention and Post-intervention
  Measures physical, psychological, social, and environmental domains of quality of life with added assessments of disability-related and autism-specific quality of life.

OTHER OUTCOMES:
Blood-oxygen-level dependent (BOLD) response in brain regions activated during a self-reflection fMRI task | Baseline; Pre-intervention
  Measure of brain activation during an fMRI task validated by Sterling (2006) requiring judgments on adjectives relating to a self-condition or judgments on whether an adjective is positively valanced.
Blood-oxygen-level dependent (BOLD) response in brain regions activated during a self-reflection fMRI task | Post-intervention (~10 weeks)
  Measure of brain activation during an fMRI task validated by Sterling (2006) requiring judgments on adjectives relating to a self-condition or judgments on whether an adjective is positively valanced.
Blood-oxygen-level dependent (BOLD) response in regions activated during an emotion-regulation fMRI task | Baseline; Pre-intervention
  Measure of brain activation during an fMRI task validated by Richey (2015) requiring regulation of emotional response to images of faces.
Blood-oxygen-level dependent (BOLD) response in regions activated during an emotion-regulation fMRI task | Post-intervention (~10 weeks)
  Measure of brain activation during an fMRI task validated by Richey (2015) requiring regulation of emotional response to images of faces.
Event-Related Potentials (ERP) measured during regulation of affective responses | Baseline; Pre-intervention
  Measure of ERP responses during an EEG task validated by Varnum (2016) requiring regulation of affective responses to both positively and negatively valenced stimuli.
Event-Related Potentials (ERP) measured during regulation of affective responses | Post-intervention (~10 weeks)
  Measure of ERP responses during an EEG task validated by Varnum (2016) requiring regulation of affective responses to both positively and negatively valenced stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany B Braden, PhD, Principal Investigator — Assistant Professor; Autism and Brain Aging Laboratory Director
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in a publication will be available upon request to approved researchers.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available upon request starting 6 months after publication and will remain available for 2 years.
Access Criteria: Data requests should be submitted to Dr. Braden at bbbraden@asu.edu and must include study aims and purpose and a detailed analysis plan describing how the data will be used. Requests will be reviewed by Dr. Braden and access to the data will be made available through a secure link to download the requested data.

REFERENCES:
- [Derived] Pagni BA, Hill E, Walsh MJM, Delaney S, Ogbeama D, Monahan L, Cook JR, Guerithault N, Dixon MV, Ballard L, Braden BB. Distinct and shared therapeutic neural mechanisms of mindfulness-based and social support stress reduction groups in adults with autism spectrum disorder. J Psychiatry Neurosci. 2023 Mar 29;48(2):E102-E114. doi: 10.1503/jpn.220159. Print 2023 Mar-Apr. PMID 36990468
- [Derived] Braden BB, Pagni BA, Monahan L, Walsh MJM, Dixon MV, Delaney S, Ballard L, Ware JE Jr. Quality of life in adults with autism spectrum disorder: influence of age, sex, and a controlled, randomized mindfulness-based stress reduction pilot intervention. Qual Life Res. 2022 May;31(5):1427-1440. doi: 10.1007/s11136-021-03013-x. Epub 2021 Oct 16. PMID 34655389